CLINICAL TRIAL: NCT02662465
Title: Oral Manifestations of Leukemia and Anticancer Treatment in Childhood
Brief Title: Oral Manifestations in Children With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Salomão Israel Monteiro Lourenço Queiroz, PhD student, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1174-3413
Record Dates: First submitted 2016-01-14; First posted 2016-01-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Mucositis
Keywords: Interventional; Treatment; Laser
MeSH Terms: conditions — Mucositis | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- mucositis grade 1, laser 660 (Experimental): Group 1 will include patients with oral mucositis grade 1. Sera used wavelength of 660nm, power 100mW and lluencia of 4 J / cm².
  Interventions: Procedure: Laser
- mucositis grade 2, laser 660 (Experimental): Group 2 included patients with oral mucositis grade 2. Sera used with a wavelength of 660nm, power 100mW and lluencia of 8 J / cm².
  Interventions: Procedure: Laser
- mucositis grade 3, laser 790 (Experimental): Group 3 included patients with oral mucositis grade 3 Sera used laser diode AsGaAl operating in continuous mode, with a wavelength of 790 nm, power of 100mW and fluency of 8 J / cm².
  Interventions: Procedure: Laser

INTERVENTIONS:
Procedure: Laser — Patients who develop oral mucositis even after the prevention, will be divided into three groups for laser sessions with the purpose of treatment of oral mucositis. The group assignment obeyed severity of oral mucositis.

SUMMARY:
Before the start of the selected chemotherapy patients will be treated preventively for oral mucositis. A group will carry out the mouthwash with chlorhexidine 0.12% twice a day for five days and another will be held to damage preventive therapy (wavelength of 660nm, power 100mW and lluencia of 4 J / cm² per point, with distance of 2cm between points located on the right buccal mucosa, left buccal mucosa, hard palate, upper lip and lower lip). Patients who develop oral mucositis even after the prevention, will be divided into three groups for laser sessions with the purpose of treatment of oral mucositis. The group assignment obeyed severity of oral mucositis. Group 1 will include patients with oral mucositis grade 1. Sera used wavelength of 660nm, power 100mW and lluencia of 4 J / cm². Group 2 included patients with oral mucositis grade 2. Sera used with a wavelength of 660nm, power 100mW and lluencia of 8 J / cm². Group 3 included patients with oral mucositis grade 3 Sera used laser diode AsGaAl operating in continuous mode, with a wavelength of 790 nm, power of 100mW and fluency of 8 J / cm².

DETAILED DESCRIPTION:
Before the start of the selected chemotherapy patients will be treated preventively for oral mucositis. A group will carry out the mouthwash with chlorhexidine 0.12% twice a day for five days and another will be held to damage preventive therapy (wavelength of 660nm, power 100mW and lluencia of 4 J / cm² per point, with distance of 2cm between points located on the right buccal mucosa, left buccal mucosa, hard palate, upper lip and lower lip). Patients who develop oral mucositis even after the prevention, will be divided into three groups for laser sessions with the purpose of treatment of oral mucositis. The group assignment obeyed severity of oral mucositis. Group 1 will include patients with oral mucositis grade 1. Sera used wavelength of 660nm, power 100mW and lluencia of 4 J / cm². Group 2 included patients with oral mucositis grade 2. Sera used with a wavelength of 660nm, power 100mW and lluencia of 8 J / cm². Group 3 included patients with oral mucositis grade 3 Sera used laser diode AsGaAl operating in continuous mode, with a wavelength of 790 nm, power of 100mW and fluency of 8 J / cm².

The assessment of oral mucositis will be held with the WHO classification: grade 0 = no mucositis; Grade I = erythema without injury; Grade II = ulcers, but can eat; Grade III = painful sores, but able to consume liquid food (nutrition), with support of analgesia; Grade IV = requires parenteral or enteral support and continuous analgesia.

The patient also conduct a self-assessment of pain by visual analog scale pain quantifying 0-10 before the laser section and after the first application.

Pediatric male or female, diagnosed with cancer who have not yet started cancer treatment, with otherwise healthy oral mucosa in the initial dental exam.

Patients who have already started treatment for cancer under radiotherapy or presenting traumatic factors (such as braces or restorations with sharp edges), or presenting ulcers in the mucosa at the initial examination.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric male or female, diagnosed with cancer who have not yet started cancer treatment, with otherwise healthy oral mucosa in the initial dental exam.

Exclusion Criteria:

* Patients who have already started treatment for cancer under radiotherapy or presenting traumatic factors (such as braces or restorations with sharp edges), or presenting ulcers in the mucosa at the initial examination.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Oral mucositis WHO classification | During the first two week evaluation
  The assessment of oral mucositis will be held with the WHO classification: grade 0 = no mucositis; Grade I = erythema without injury; Grade II = ulcers, but can eat; Grade III = painful sores, but able to consume liquid food (nutrition), with support of analgesia; Grade IV = requires parenteral or enteral support and continuous analgesia.

SECONDARY OUTCOMES:
Visual analog scale | A week before and week after the laser application
  The patient also conduct a self-assessment of pain by visual analog scale pain quantifying 0-10 before the laser section and after the first application.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No